CLINICAL TRIAL: NCT03200405
Title: Morphological Imaging of Meshes in Underlay Position After Treatment of Primary Umbilical Hernias: a Randomised Controlled Trial
Brief Title: Visible vs. Non-Visible Mesh in Underlay Positon After Repair of Umbilical Hernias
Acronym: NANEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Ulrich Dietz, Prof., Wuerzburg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dietz_87/16-sc
Record Dates: First submitted 2017-05-23; First posted 2017-06-27 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Umbilical Hernia
Keywords: umbilical hernia; mesh repair; MRI-visibility; underlay; NANEP; DynaMeshCICAT; DynaMeshVisible; preperitoneal
MeSH Terms: conditions — Hernia, Umbilical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DynaMeshVisible (Experimental): the umbilical hernia will be fixed with a mesh, which is incorporated with Fe3O4 particles to become visible in MRI
  Interventions: Device: DynaMeshVisible
- DynaMeshCICAT (Active Comparator): the umbilical hernia will be fixed with a Non-MRI-visible PVDF Mesh
  Interventions: Device: DynaMeshCICAT

INTERVENTIONS:
Device: DynaMeshVisible — The umbilical hernias will be fixed with a mesh. In this group a MRI-visible mesh will be used.
  Arms: DynaMeshVisible
Device: DynaMeshCICAT — The umbilical hernias will be fixed with a mesh. In this group a non-visible mesh will be used.
  Arms: DynaMeshCICAT

SUMMARY:
The purpose of this study is to determine the exact position of a mesh which is placed in underlay position in umbilical hernia in vitro. The investigators want to gain information if the mesh lays directly next to the abdominal wall fascia or if there´s fat tissue between mesh and fascia. Furthermore they hope to get some information about the tissue incorporation.

DETAILED DESCRIPTION:
The literature tells to supply umbilical hernia with a mesh, that overlaps 5-6 cm in each direction. To achieve this overlap an extensive taxidermy is necessary, which causes a big operation trauma. An umbilical hernia is an extended physiological stoma and compared to an incisional hernia has no risk to rip further. Therefore the researchers act on the assumption that this generous overlap is not necessary. For a short time there is a new mesh available, which combines all the necessary requirements as elasticity, effective porousness and a structure of monofilaments with MRI visibility. In a randomised clinical trial two sorts of meshes, a conventional PVDF(polyvinylidene fluoride) mesh (DynaMesh-CICAT) and a MRI visible PVDF(polyvinylidene fluoride) mesh (DynaMeshVisible) shall be compared.The investigators postulate that there is no difference between the two groups concerning complications, relapse and life quality after 4 weeks and 12 months. Altogether the goal of the study is to determine the exact position of the mesh in vitro.

The study design is a double-blinded, multicentric randomised controlled study. The radiologist and the examiner are blinded. It will be reported according to the CONSORT Statements.

The eligibility criteria is written anywhere else. The operation results after an single shot antibiotics in open method. The access happens via a semicircular infraumbilical cut. There will be prepared until the linea alba and the umbilical hernia orifice to display the hernia gap and the hernia sac. If there´s only a fat prolapse, it will be removed by ligation. If there´s an peritoneal hernia sac, the content will be repositioned and the hernia sac will be removed. The preperitoneal space will be prepared bluntly and the peritoneum will be released from the rectus sheath. A 4-6 cm trimmed mesh with a central thread will be inserted in underlay position. The central thread is used for orientation. The hernial gap will be closed in transversal direction with absorbable threads. After the reinsertion of the navel the region of the operation will be closed with subcutaneous und intracutaneous seams.

The randomisation succeeded via block randomisation at a ratio of 1 to 1. A randomisation list with SAS®-Makros "Randomisation Tables" by M. Stout is already created. There is one list for Wuerzburg and one for Kitzingen. In total there are 72 assignments created, instead of 50. But upon consultation the recruitment will be stopped after the 50th patient. According to the calculations of the epidemiological departement of the University of Wuerzburg there are 22 patients needed in each arm, that means 44 patients in total to reach the confidence interval. The patient data will be imported to EuraHS. This data entry is based on the ethics committee vote of the medical departement of Wuerzburg dated the 31th of july 2012 (application number 256/11) and the renewal of the 21st of july 2015.

If there´s an increased complication rate in one of the groups or the morphology of the MRI-visible meshes is found unsatisfactory the study will be cancelled.

The patient data will be recorded via pseudonyms.

ELIGIBILITY:
Inclusion Criteria:

* umbilical hernia > 0,4 cm; <= 3 cm
* BMI > 20; < 51

Exclusion Criteria:

* emergency operation
* previous abdominal operation
* epigastric hernia in more than 3 cm distance of the umbilical hernia
* ascites
* hepatic insufficiency
* periumbilical skin disease
* incisional umbilical hernia
* claustrophobia
* contraindications concerning the MRI examination

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
MRI visibility and visible size of the mesh 4 weeks after operation | 4 weeks
  A MRI will be done 4 weeks after the operation and it will be registered if the mesh is visible; furthermore there will be done some measurements to specify the exact position and the visible size of the mesh

SECONDARY OUTCOMES:
MRI visibility and visible size of the mesh 12 months after operation | 12 months
  A MRI will be done 12 months after the operation and it will be registered if the mesh is visible; furthermore there will be done some measurements to specify the exact position and the visible size of the mesh
intraoperative and postoperative complications (30-day morbidity) | 4 weeks
  There will be registered if there are any intraoperative or postoperative complications
relapse 12 months after operation | 12 months
  There will be registered if there is an relapse 12 months after operation.
life quality 4 weeks and 12 months after operation | 12 months
  There will be done a questionnaire 4 weeks and 12 months after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Dietz, Prof Dr Dr, Principal Investigator — Wuerzburg UH
Locations (1):
- Universitätsklinikum Wuerzburg, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No